CLINICAL TRIAL: NCT02980055
Title: Comparison of Root Coverage of Gingival Recessions Using Connective Tissue Graft and Collagen Matrix
Brief Title: Comparison of Root Coverage of Gingival Recessions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Karyna de Melo Menezes, Principal Invastigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFRN-3
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Gingival Recession
Keywords: connective tissue graft; transplantation; collagen; autologous; gingiva
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test: collagen matrix (Experimental): Root coverage using collagen matrix
  Interventions: Procedure: collagen matrix
- Control: connective tissue graft (Active Comparator): Root coverage using connective tissue graft
  Interventions: Procedure: connective tissue graft

INTERVENTIONS:
Procedure: collagen matrix — Surgical procedure for root coverage using collagen matrix
  Other Names: xenogeneic collagen matrix
  Arms: Test: collagen matrix
Procedure: connective tissue graft — Surgical procedure for root coverage using connective tissue graft
  Other Names: autologous
  Arms: Control: connective tissue graft

SUMMARY:
The purpose of this study is to analyze the percentage of root coverage in Miller class I and II gingival recessions using connective tissue graft and collagen matrix with a two years follow-up.

DETAILED DESCRIPTION:
A sample calculation using a mean of 2.92 mm of the quantity of keratinized mucosa obtained after six months in the most recent study (McGUIRE; SCHEYER, 2014) using the same collagen matrix with a standard deviation of ± 0.88 mm, a difference of 0.4 mm being chosen as statistically significant. In addition, a 95% bilateral confidence interval and 80% power were used. A sample of 38 individuals per group was obtained. In addition, a 20% loss is expected during follow-up, a total of 46 individuals should be evaluated.

Periapical radiographic examinations should be performed before the collection of data to confirm the absence of bone loss. The following clinical parameters should be evaluated in both test and control groups: visible plaque index, gingival bleeding index, gingival recession, keratinized mucosa width and thickness, probing depth, bleeding on probing and periodontal biotype for each teeth with a North Carolina periodontal probe. The periodontal biotype for each teeth should be rated as thin or thick, according to probe transparency during probing depth. For statistical purposes, percentages of faces with gingival recession should be calculated. These parameters should be evaluated at baseline and at one, three and six months, one and two years post-therapy.

Clinical parameters should be collected by two operators, calibrated by the Kappa test for the keratinized mucosa width and thickness, periodontal biotype, probing depth and gingival recession.

After the inclusion of the patients, anamnesis and initial examination were performed. The subjects should be divided randomly, using a simple draw, in the following two groups: test - (collagen matrix) and control - (connective tissue graft) placebo associated with basic periodontal therapy). The data should be analyzed using descriptive and inferential statistics, with parametric tests, through the software package Social Sciences (SPSS), version 17.0 (free version).

ELIGIBILITY:
Inclusion Criteria:

* Gingival recessions of class I or II types according to Miller (1985), in contralateral, superior or inferior premolars and / or canines;
* Fine periodontal biotype characterized by the transparency of the North Carolina probe when introduced into the periodontal sulcus (KAN et al., 2003);
* The teeth with gingival recession should not be restored in their cervical portion;
* Periodontal health characterized by absence of bleeding at probing, depth of probing less than 3 mm;
* Visible Plaque Index and Gingival Bleeding Index less than or equal to 30%.

Exclusion Criteria:

* Orthodontic appliances;
* Fixed or removable prostheses involving the premolar teeth with gingival recession;
* Being a smoker;
* Pregnancy or lactation;
* Systemic diseases that may interfere with healing or periodontal health (diabetes, leukemia, hypertension, among others).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
gingival recession | baseline
gingival recession | three months
gingival recession | six months
gingival recession | twelve months
gingival recession | eighteen months
gingival recession | twenty-four months

SECONDARY OUTCOMES:
Width of keratinized mucosa | baseline and three, six, twelve, eighteen and twenty-four months

CONTACTS AND LOCATIONS:
Overall Officials: Karyna M Menezes, Master, Principal Investigator — Universidade Federal do Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No